CLINICAL TRIAL: NCT05277688
Title: Adjuvant Concurrent Chemoradiotherapy Versus Radiotherapy in Early-stage Cervical Cancer Patients With Selected Intermediate-risk Factors: a Randomized Controlled Phase III Trials (ACCEPT Trial)
Brief Title: Adjuvant Concurrent Chemoradiotherapy Versus Radiotherapy in Early-stage Cervical Cancer Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021(237)
Record Dates: First submitted 2022-03-02; First posted 2022-03-14 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-03

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; early stage; chemoradiotherapy; radiotherapy; survival
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): concurrent chemotherapy: cisplatin（DDP） weekly, 40mg/m2, begin with radiation Drug: cisplatin（DDP） weekly; pelvic radiotherapy: intensity modulated radiotherapy (IMRT) is given five fractions per week at 1.8-2 Gy/fraction/day with total dose summed up to 45-50Gy.
  Interventions: Drug: adjuvant concurrent chemoradiotherapy
- controlled group (Active Comparator): pelvic radiotherapy alone: intensity modulated radiotherapy (IMRT) is given five fractions per week at 1.8-2 Gy/fraction/day with total dose summed up to 45-50Gy.
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Drug: adjuvant concurrent chemoradiotherapy — concurrent chemotherapy: cisplatin（DDP） weekly, 40mg/m2, begin with radiation Drug: cisplatin（DDP） weekly; Intensity modulated radiotherapy (IMRT) is given five fractions per week at 1.8-2 Gy/fraction/day with total dose summed up to 45-50Gy.
  Arms: experimental group
Radiation: radiotherapy — Intensity modulated radiotherapy (IMRT) is given five fractions per week at 1.8-2 Gy/fraction/day with total dose summed up to 45-50Gy.
  Arms: controlled group

SUMMARY:
To evaluate if adjuvant concurrent chemoradiotherapy is associated with a recurrence-free survival benefit in comparison with radiotherapy alone in selected intermediate risk cervical cancer after radical surgery.

DETAILED DESCRIPTION:
Adjuvant therapy for patients with cervical cancer (CC) with intermediate-risk factors remains controversial. According to result of GOG 92 trail, adjuvant radiotherapy significantly improved recurrence-free survival in early stage cervical cancer with intermediate risks (Sedlis criteria). However, significant heterogeneity exists in Sedlis criteria, high risk of relapse and death occurred in patients with (1) lympho-vascular space invasion(LVSI+) and deep 1/3 stromal invasion;(2) LVSI(+) and middle 1/3 stromal invasion, and tumor size≥4cm when compared with other factors. In addition, multiple studies have confirmed that (3)non-squamous histology is an independent prognostic factor in early stage cervical cancer, who might be benefited from adjuvant concurrent chemoradiotherapy. As a result, The objective of the trial is to evaluate if adjuvant concurrent chemoradiotherapy is associated with a recurrence-free survival benefit in comparison with radiotherapy alone in selected intermediate risk cervical cancer after radical surgery. The primary endpoint of the study is the recurrence-free survival from the day of randomization.

ELIGIBILITY:
Inclusion Criteria:

* • 18 Years to 80 Years

  * Histologically proven cervical cancer, FIGO stage Ia2-IIb,and no previous chemotherapy and radiotherapy
  * Accepted radical hysterectomy 3-4 weeks before
  * Karnofsky score >70
  * Postoperative pathology with one of the three risk factors criterials: (1) lympho-vascular space invasion(LVSI+) and deep 1/3 stromal invasion; (2 ) LVSI(+) and middle 1/3 stromal invasion, and tumor size≥4cm (3)Non-squamous cell carcinoma;
  * Examination results showed no radiation or chemotherapy contraindication
  * Willing to accept treatment
  * Ability to comply with trial requirements

Exclusion Criteria:

* • Postoperative residual

  * Postoperative recurrence or metastasis
  * Pelvic lymph node metastasis
  * parametrial invasion
  * positive surgical margin
  * Without lymph node dissection
  * Postoperative pathology showed aortic lymph node metastasis
  * Examination results showed radiotherapy contraindications
  * No indications for radiotherapy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — cervical cancer is only found and diagnosed in female patients
Enrollment: 340 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
5-year recurrence-free survival | 5 years
  From date of surgery until the date of first documented local-regional progression or distant metastasis (determined by CT or MRI scan and/or biopsy) or death (from any cause) assessed up to five years.

SECONDARY OUTCOMES:
5-year overall survival | 5 years
  Determine the 5-year overall survival rate in early-stage cervical cancer patients with high risk factors, defined as time from the date of surgery to death of all cause at time of 5 years after operation.
Acute toxicity | 3 months
  Evaluate the treatment induced toxicity according to CTCAE 4.0 during the time of chemoradiotherapy or radiotherapy alone which starts from the first day of Endostar and lasts three months.
Quality of Life (QoL) | 2 years
  Collect QoL data on early-stage cervical cancer patients with high risk factors. The data is measured by EORTC QLQ-C30 (Version 3.0) according to investigator collection at the starting and ending time of the adjuvant treatment. EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients. The core and disease-specific for cervix modules are selected to estimate treatment related influence on patients' life. The final score of the questionnaire is collected and analyzed according to detailed scoring procedures from manuals.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai jiaotong univestigy school of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
we donot plan to share the IPD data about the trial